CLINICAL TRIAL: NCT03977727
Title: An Exploratory, Single-center, Randomized, Open Label, Active-control, Cross-over Trial Comparing the Efficacy and Safety of Continuous Subcutaneous Insulin Infusion of Faster-acting Insulin Aspart (Fiasp®) Compared to NovoLog® Used in the Medtronic 670G Closed Loop System in Adults With Type 1 Diabetes
Brief Title: FIasp® vs. Novolog® in Type 1 Diabetics Using 670G Medtronic Pump
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Texas Diabetes & Endocrinology, P.A. (Other)
Responsible Party: Principal Investigator, Thomas C. Blevins, M.D., PI, Texas Diabetes & Endocrinology, P.A.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: U1111-1213-9104
Record Dates: First submitted 2019-04-17; First posted 2019-06-06 (Actual); Results first posted 2020-09-09 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-08

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Fiasp/Novolog (Experimental): 7 weeks on Fiasp® then crossover to 7 weeks on Novolog® in subjects on the 670g Hybrid Closed Loop Continuous Subcutaneous Insulin Infusion
  Interventions: Drug: Fiasp®; Drug: Novolog®; Device: 670G hybrid closed loop continuous subcutaneous insulin infusion system
- Novolog/Fiasp (Experimental): 7 weeks on Novolog® then crossover to 7 weeks on Fiasp® in subjects on the 670g Hybrid Closed Loop Continuous Subcutaneous Insulin Infusion
  Interventions: Drug: Fiasp®; Drug: Novolog®; Device: 670G hybrid closed loop continuous subcutaneous insulin infusion system

INTERVENTIONS:
Drug: Fiasp® — Fiasp® used in a 670G hybrid closed loop continuous subcutaneous insulin infusion system
Drug: Novolog® — Novolog® used in a 670G hybrid closed loop continuous subcutaneous insulin infusion system
  Other Names: Aspart
Device: 670G hybrid closed loop continuous subcutaneous insulin infusion system — CSII
  Other Names: Medtronic 670G pump

SUMMARY:
This is an exploratory, single-center, randomized, open label, active-controlled, complete cross-over trial comparing safety and efficacy of Fiasp® versus NovoLog® when used in the Medtronic MiniMed 670G system in subjects with T1DM.

DETAILED DESCRIPTION:
This study is being performed to compare Fiasp® in terms of glycemic control with a focus on post-prandial 1-hour plasma glucose level and system-based outcomes to NovoLog® insulin when used in the Medtronic mini Med 670G HCL system (operating in auto-mode) in patients with type 1 diabetes. The investigator's hypothesis is that post prandial glucoses will be lower and time in range will be greater during the Fiasp® treatment period.

Subjects will have a 2 week screening period, 14 week treatment period and 30 Day follow up period. After at least 7 weeks on treatment period one they will crossover to treatment period two on the opposite treatment for 7 additional weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent obtained before any trial-related activities. Trial-related activities are any procedures that are carried out as part of the trial, including activities to determine suitability for the trial
2. Male or female, age ≥18 years at the time of signing informed consent
3. Documented diagnoses of T1DM ≥1 year prior to the day of screening
4. Using the Medtronic pump Minimed 670G for CSII in a basal-bolus regimen with a rapid acting insulin analogue for at least 30 days prior to screening and willing to continue using their personal Medtronic Minimed 670G and CSII for insulin treatment throughout the trial.
5. Ability and willingness to use the same insulin infusion sets throughout the trial
6. Using the same insulin for at least 30 days prior to screening
7. HbA1c < 8.5% as assessed by local laboratory at screening
8. BMI ≤ 35.0 kg/m2 at screening
9. Ability and willingness to adhere to the protocol including performing SMPG profiles, attending visits, utilizing the auto mode feature of the pump for at least 80 % of the time during the study, and completing meal tests

Exclusion Criteria:

1. Known or suspected hypersensitivity to trial products or related products
2. Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using adequate contraceptive methods (adequate contraceptive measures as required by local regulation or practice)
3. Participation in another clinical trial within 28 days before the screening visit. Note: clinical trials do not include non-interventional studies
4. Anticipated significant change in lifestyle (e.g. eating, exercise or sleeping pattern) throughout the trial
5. Any of the following: myocardial infarction, stroke, hospitalization for unstable angina or transient ischemic attack within the past 180 days prior to the day of screening
6. Subjects classified as being in New York Heart Association (NYHA) Class IV at screening
7. Planned coronary, carotid or peripheral artery revascularization known on the day of screening.
8. Inadequately treated blood pressure defined as Grade 3 hypertension or higher (Systolic

   ≥180 mmHg or diastolic ≥110 mmHg) at screening
9. Impaired liver function, defined as ALT ≥ 2.5 times upper normal limit at screening
10. Renal impairment measured as estimated Glomerular Filtration Rate (eGFR) value of < 45 ml/min/1.73 m2
11. Anticipated initiation or change in concomitant medications (for more than 14 consecutive days) known to affect weight or glucose metabolism in the opinion of the Investigator
12. Proliferative retinopathy or maculopathy requiring acute treatment at the time of screening
13. History of hospitalization for ketoacidosis ≤180 days prior to the day of screening
14. Treatment with any medication for the indication of diabetes or obesity other than stated in the inclusion criteria within 30 days before screening
15. Presence of malignant neoplasms at the time of screening. Basal and squamous cell skin cancer and any carcinoma in-situ is allowed.
16. Reoccurring Severe hypoglycemia while on the Medtronic Minimed 670G in the investigators opinion
17. Any condition which, in the opinion of the Investigator, might jeopardize Subject's safety or compliance with the protocol

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-06-11 (Actual); Primary Completion 2020-03-09 (Actual); Study Completion 2020-04-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Blevins, MD, Principal Investigator — Texas Diabetes & Endocrinology
Locations (1):
- Texas Diabetes & Endocrinology, Austin, Texas, United States

REFERENCES:
- [Derived] Ozer K, Cooper AM, Ahn LP, Waggonner CR, Blevins TC. Fast Acting Insulin Aspart Compared with Insulin Aspart in the Medtronic 670G Hybrid Closed Loop System in Type 1 Diabetes: An Open Label Crossover Study. Diabetes Technol Ther. 2021 Apr;23(4):286-292. doi: 10.1089/dia.2020.0500. Epub 2021 Mar 8. PMID 33090016

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 45 patients were screened for eligibility between June 11,2019 and November 21, 2019 at a diabetes clinic in Austin, TX
Pre-assignment Details: 40 of 45 participants were randomized. All 5 who were not randomized did not meet inclusion criteria.
Period: First Treatment
Arm/Group | Fiasp/Novolog | Novolog/Fiasp
Started | 20 | 20
Received Treatment | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0
Period: Second Treatment
Arm/Group | Fiasp/Novolog | Novolog/Fiasp
Started | 20 | 20
Completed | 20 | 17
Not Completed | 0 | 3
Not completed — Lost to Follow-up | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fiasp/Novolog | Novolog/Fiasp | Total
Number analyzed (Participants) | 20 | 17 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.2 (13.17) | 43.8 (12.77) | 45.7 (27.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 4 | 12
  Male | 12 | 13 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 19 | 16 | 35
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 20 | 17 | 37
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 17 | 37
BMI [Mean (Standard Deviation); unit: kg/m^2] | 26.9 (3.69) | 27.3 (3.15) | 27.1 (3.41)
Weight [Mean (Standard Deviation); unit: kg] | 80.3 (14.7) | 83.3 (12.45) | 81.7 (13.61)
Height [Mean (Standard Deviation); unit: cm] | 172.3 (10.82) | 174.6 (7.22) | 173.4 (9.29)

OUTCOME MEASURES:

1. Primary Outcome: 1-Hour Change in Postprandial Plasma Glucose (PPG)
Description: Change was calculated as the PPG value at 1 hour minus the PPG value at baseline (time -2 minutes) during meal test
Time Frame: 6th week of therapy
Population: All patients who participated in the meal test after 6 weeks of therapy in each arm
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- Fiasp/Novolog: Participants with type 1 diabetes spent 6 weeks on Fiasp® then crossed over to 6 weeks on Novolog®
- Novolog/Fiasp: Participants with type 1 diabetes spent 6 weeks on Novolog® then crossed over to 6 weeks on Fiasp®
Arm/Group | Fiasp/Novolog | Novolog/Fiasp
Number analyzed (Participants) | 20 | 17
mg/dL
  Fiasp | 105.15 (56.73) | 154.24 (54.25)
  NovoLog | 99.90 (82.70) | 114.94 (61.14)
Statistical Analysis 1: Comparison: Fiasp/Novolog vs Novolog/Fiasp; Linear mixed model was fit with therapy (Fiasp vs. NovoLog), period (Period 1 vs Period 2), and sequence (Fiasp/NovoLog vs NovoLog/Fiasp) as fixed effects. Subjects included as random effects; Test type: Superiority; p = .008, Mixed Models Analysis; Mean Difference (Final Values) = 27.35, 95% CI 2-sided [7.88 to 48.4]

2. Secondary Outcome: 2-Hour Change in Postprandial Plasma Glucose (PPG)
Description: Change was calculated as the value at 2 hour minus the value at baseline during meal test
Time Frame: 6th week of therapy
Population: All patients who participated in the meal test after 6 weeks of therapy in each arm
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Fiasp/Novolog | Novolog/Fiasp
Number analyzed (Participants) | 20 | 17
mg/dL
  Fiasp | 72.55 (90.62) | 65.00 (57.22)
  NovoLog | 69.10 (92.55) | 104.53 (80.57)
Statistical Analysis 1: Comparison: Fiasp/Novolog vs Novolog/Fiasp; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .136, Mixed Models Analysis; Mean Difference (Final Values) = 15.22, 95% CI 2-sided [-5.42 to 39.46]

3. Secondary Outcome: Percentage of Time Spent Between Below 70 mg/dL
Description: Percent of time spent is calculated as the accumulated time in hours spent within each range divided by the total number of hours spent under therapy with each drug (6 weeks each)
Time Frame: Weeks 1 through 6, Weeks 8 through 13
Population: All patients for whom continuous glucose monitoring data was available during the specified time periods
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Fiasp/Novolog | Novolog/Fiasp
Number analyzed (Participants) | 20 | 17
percentage of time
  Fiasp | 1.94 (1.48) | 1.72 (1.20)
  NovoLog | 2.42 (1.62) | 2.03 (1.36)
Statistical Analysis 1: Comparison: Fiasp/Novolog vs Novolog/Fiasp; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .029, Mixed Models Analysis; Mean Difference (Final Values) = .4, 95% CI 2-sided [.05 to .73]

4. Secondary Outcome: Percentage of Time Spent Between 70 mg/dL and 180 mg/dL
Description: as for outcome 3
Time Frame: Weeks 1 through 6, Weeks 8 through 13
Population: All patients for whom continuous glucose monitoring data was available during the specified time periods
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Fiasp/Novolog | Novolog/Fiasp
Number analyzed (Participants) | 20 | 17
percentage of time
  Fiasp | 74.80 (8.08) | 73.67 (6.80)
  NovoLog | 70.28 (8.12) | 75.04 (5.95)
Statistical Analysis 1: Comparison: Fiasp/Novolog vs Novolog/Fiasp; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .016, Mixed Models Analysis; Mean Difference (Final Values) = -1.81, 95% CI 2-sided [-2.84 to -0.31]

5. Secondary Outcome: Percentage of Time Spent Above 200 mg/dL
Description: as for outcome 3
Time Frame: Weeks 1 through 6, Weeks 8 through 13
Population: All patients for whom continuous glucose monitoring data was available during the specified time periods
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Fiasp/Novolog | Novolog/Fiasp
Number analyzed (Participants) | 20 | 17
percentage of time
  Fiasp | 14.90 (6.90) | 15.44 (5.65)
  NovoLog | 18.57 (7.85) | 14.11 (4.43)
Statistical Analysis 1: Comparison: Fiasp/Novolog vs Novolog/Fiasp; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .045, Mixed Models Analysis; Mean Difference (Final Values) = 1.38, 95% CI 2-sided [.04 to 2.32]

6. Secondary Outcome: Percentage of Time Spent in Hypoglycemia (40 mg/dL - 54 mg/dL)
Description: as for outcome 3
Time Frame: Weeks 1 through 6, Weeks 8 through 13
Population: All patients for whom continuous glucose monitoring data was available during the specified time periods
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Fiasp/Novolog | Novolog/Fiasp
Number analyzed (Participants) | 20 | 17
percentage of time
  Fiasp | .46 (.53) | .40 (.48)
  NovoLog | .50 (.50) | .35 (.36)

7. Secondary Outcome: Percentage of Time Spent in Severe Hypoglycemia (> 40 mg/dL)
Description: as for outcome 3
Time Frame: Weeks 1 through 6, Weeks 8 through 13
Population: All patients for whom continuous glucose monitoring data was available during the specified time periods
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Fiasp/Novolog | Novolog/Fiasp
Number analyzed (Participants) | 20 | 17
percentage of time
  Fiasp | 0 (0) | 0 (0)
  NovoLog | 0 (0) | 0 (0)

8. Secondary Outcome: 1,5 Anhydroglucitol Levels
Description: 1,5 anhydroglucitol levels were measured on the 6th week of each therapy
Time Frame: Week 6, Week 13
Population: All patients who participated in the meal test after 6 weeks of therapy in each period
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Fiasp/Novolog | Novolog/Fiasp
Number analyzed (Participants) | 20 | 17
µg/mL
  Fiasp | 6.50 (3.37) | 7.12 (3.23)
  NovoLog | 6.28 (3.54) | 6.95 (3.31)
Statistical Analysis 1: Comparison: Fiasp/Novolog vs Novolog/Fiasp; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .303, Mixed Models Analysis; Mean Difference (Final Values) = -.2, 95% CI 2-sided [-.59 to .16]

9. Secondary Outcome: Fructosamine Levels
Description: Cumulative glycemic control expressed in fructosamine levels (micromol/Liter) were measured on the 6th week of each therapy
Time Frame: Week 6, Week 13
Population: All patients who participated in the meal test after 6 weeks of therapy in each period
Measure: Mean (Standard Deviation); unit: mcmol/L
Arm/Group | Fiasp/Novolog | Novolog/Fiasp
Number analyzed (Participants) | 20 | 17
mcmol/L
  Fiasp | 322.60 (42.24) | 296.35 (31.10)
  NovoLog | 305.40 (32.28) | 314.31 (28.97)
Statistical Analysis 1: Comparison: Fiasp/Novolog vs Novolog/Fiasp; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .968, Mixed Models Analysis; Mean Difference (Final Values) = -1.18, 95% CI 2-sided [-10.32 to 9.99]

10. Secondary Outcome: HbA1c
Description: Cumulative glycemic control expressed in HbA1c% measured on the 6th week of each therapy
Time Frame: Week 6, Week 13
Population: All patients who participated in the meal test after 6 weeks of therapy in each period
Measure: Mean (Standard Deviation); unit: HbA1c%
Arm/Group | Fiasp/Novolog | Novolog/Fiasp
Number analyzed (Participants) | 20 | 17
HbA1c%
  Fiasp | 7.09 (.47) | 7.00 (.31)
  NovoLog | 7.09 (.44) | 6.88 (.33)
Statistical Analysis 1: Comparison: Fiasp/Novolog vs Novolog/Fiasp; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .059, Mixed Models Analysis; Mean Difference (Final Values) = -.06, 95% CI 2-sided [-.13 to 0]

11. Secondary Outcome: Insulin Use - Change in Daily Dose
Description: Change was calculated as the value on the last day of therapy minus the value on the 1st day of therapy in each period
Time Frame: Weeks 1 through 6, Weeks 8 through 13
Population: All patients who participated in the meal test after 6 weeks of therapy in each arm
Measure: Mean (Standard Deviation); unit: units
Arm/Group | Fiasp/Novolog | Novolog/Fiasp
Number analyzed (Participants) | 20 | 17
units
  Fiasp | -2.1 (7.45) | .29 (13.35)
  NovoLog | 1.10 (11.80) | -2.65 (9.13)

12. Secondary Outcome: Insulin Use - Bolus
Description: Change in %bolus insulin (units) as the value on the last day of therapy minus the value on the 1st day of therapy in each period
Time Frame: Weeks 1 through 6, Weeks 8 through 13
Population: All patients who participated in the meal test after 6 weeks of therapy in each arm
Measure: Mean (Standard Deviation); unit: percentage of units
Arm/Group | Fiasp/Novolog | Novolog/Fiasp
Number analyzed (Participants) | 20 | 17
percentage of units
  Fiasp | -1.54 (6.54) | -4.32 (7.85)
  NovoLog | 1.83 (7.62) | -1.34 (5.35)

13. Secondary Outcome: Insulin Use - Basal
Description: Change in %basal insulin (units) as the value on the last day of therapy minus the value on the 1st day of therapy in each period
Time Frame: Weeks 1 through 6, Weeks 8 through 13
Population: All patients who participated in the meal test after 6 weeks of therapy in each arm
Measure: Mean (Standard Deviation); unit: percentage of units
Arm/Group | Fiasp/Novolog | Novolog/Fiasp
Number analyzed (Participants) | 20 | 17
percentage of units
  Fiasp | 1.54 (6.54) | 4.32 (7.85)
  NovoLog | -1.83 (7.62) | 1.34 (5.35)

14. Secondary Outcome: Insulin Use - Automatic Basal Insulin
Description: Average amount per day (units) calculated for each participant under each therapy
Time Frame: Weeks 1 through 6, Weeks 8 through 13
Population: All patients who participated in the meal test after 6 weeks of therapy in each arm
Measure: Mean (Standard Deviation); unit: units
Arm/Group | Fiasp/Novolog | Novolog/Fiasp
Number analyzed (Participants) | 20 | 17
units
  Fiasp | .87 (.307) | 1.20 (.65)
  NovoLog | .86 (.32) | 1.20 (.66)

15. Secondary Outcome: Insulin Pump - Active Insulin Time
Description: Average time per day (hours) calculated for each participant under each therapy
Time Frame: Weeks 1 through 6, Weeks 8 through 13
Population: All patients who participated in the meal test after 6 weeks of therapy in each arm
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Fiasp/Novolog | Novolog/Fiasp
Number analyzed (Participants) | 20 | 17
hours
  Fiasp | 3 (.06) | 3 (0)
  NovoLog | 3 (0) | 3 (.02)

16. Secondary Outcome: Insulin Pump - Auto Mode
Description: Percentage of time spent in auto-mode after calibration under each therapy
Time Frame: Weeks 3 through 6, Weeks 10 through 13
Population: All patients who participated in the meal test after 6 weeks of therapy in each arm
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Fiasp/Novolog | Novolog/Fiasp
Number analyzed (Participants) | 20 | 17
percentage of time
  Fiasp | 89.28 (6.42) | 89.31 (8.42)
  NovoLog | 86.17 (11.43) | 87.2 (15.6)

17. Secondary Outcome: Insulin Pump - Manual Mode
Description: Percentage of time spent in manual-mode after calibration under each therapy
Time Frame: Weeks 3 through 6, Weeks 10 through 13
Population: All patients who participated in the meal test after 6 weeks of therapy in each arm
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Fiasp/Novolog | Novolog/Fiasp
Number analyzed (Participants) | 20 | 17
percentage of time
  Fiasp | 10.72 (6.42) | 10.69 (8.42)
  NovoLog | 13.45 (11.44) | 12.8 (15.6)

18. Secondary Outcome: Change in Carbohydrate Ratio
Description: Change was calculated as the carbohydrate ratio on the last day of therapy minus the carbohydrate ratio on the 1st day of therapy in each period
Time Frame: Weeks 1 through 6, Weeks 8 through 13
Population: All patients who participated in the meal test after 6 weeks of therapy in each arm
Measure: Mean (Standard Deviation); unit: I:CR
Arm/Group | Fiasp/Novolog | Novolog/Fiasp
Number analyzed (Participants) | 20 | 17
I:CR
  Fiasp | -.27 (1.09) | -.02 (.47)
  NovoLog | -.14 (.95) | .2 (.76)

19. Secondary Outcome: Infusion Site Reactions
Description: Number of Infusion site reactions reported by patient
Time Frame: 14 week treatment period
Population: All patients who participated in the meal test after 6 weeks of therapy in each arm
Measure: Number; unit: occurances
Arm/Group | Fiasp/Novolog | Novolog/Fiasp
Number analyzed (Participants) | 20 | 17
occurances
  Fiasp | 0 | 1
  NovoLog | 3 | 2

20. Secondary Outcome: Pump Occlusions
Description: Number of Occlusion events reported by patient
Time Frame: 14 week treatment period
Population: All patients who participated in the meal test after 6 weeks of therapy in each arm
Measure: Number; unit: occurances
Arm/Group | Fiasp/Novolog | Novolog/Fiasp
Number analyzed (Participants) | 20 | 17
occurances
  Fiasp | 7 | 6
  NovoLog | 7 | 9

ADVERSE EVENTS:
Time Frame: Approximately 20 weeks. The entire duration of the subjects study period.
Description: Adverse event information was collected at all phone or office visits during the trial.
Arm/Group | Fiasp/Novolog | Novolog/Fiasp
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/18
Serious Adverse Events (participants affected / at risk) | 1/19 | 0/18
Other Adverse Events (participants affected / at risk) | 11/19 | 7/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fiasp/Novolog (N=19) | Novolog/Fiasp (N=18)
Herniated Disc (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Subject hospitalized for laminectomy to repair herniated disc
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fiasp/Novolog (N=19) | Novolog/Fiasp (N=18)
Non Proliferative Diabetic Retinopathy (Eye disorders) | 0 (0) | 1 (1)
Worsening of Seasonal Allergic Rhinitis (General disorders) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Redness at infusion site (right abdomen) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Trivial tricuspid regurgitation (Cardiac disorders) | 0 (0) | 1 (18)
Trivial mitral regurgitation (Cardiac disorders) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Sore Throat (General disorders) | 0 (0) | 1 (1)
Headache (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal Congestion (General disorders) | 0 (0) | 1 (1)
First Degree AV Block (Cardiac disorders) | 0 (0) | 1 (1)
Intermittent Heart Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Intermittent bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Worsening of Hypertension (Cardiac disorders) | 1 (1) | 0 (0)
Conjuntivitis (Infections and infestations) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 1 (1)
Gasteroenteritis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Supraventricular Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Herniated Disc (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Abdominal Cramps (General disorders) | 1 (1) | 0 (0)
Emesis (General disorders) | 1 (1) | 0 (0)
Traveler's Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hiatial Hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Irritation at Infusion site (abdoment) (Product Issues) | 0 (0) | 1 (1) — related to infusion site , not insulin
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Right Thumb laceration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Common Cold (Infections and infestations) | 2 (3) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Worsening of hypocalcemia (Endocrine disorders) | 0 (0) | 1 (1)
erythema at infusion site (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Sinus Infection (Infections and infestations) | 0 (0) | 1 (1)
Right index finger dislocation (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Triangular fibrocartilage band tear (left wrist) (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Worsening of hypothyroidsm (Endocrine disorders) | 1 (1) | 0 (0)
myalgia (bilateral shoulders0 (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Ecchymosis (bilateral hands) (General disorders) | 1 (1) | 0 (0)
acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Hyperkalemia (Cardiac disorders) | 1 (1) | 0 (0)
Center involved diabetic macular edema (right eye) (Eye disorders) | 1 (1) | 0 (0)
Vasovagal Syncope (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-16): https://cdn.clinicaltrials.gov/large-docs/27/NCT03977727/Prot_SAP_000.pdf